CLINICAL TRIAL: NCT00460967
Title: Safety and Effectiveness, in a Multi-Center, Randomized, Sham Controlled Investigation for Dry, Non-Exudative Age Related Macular Degeneration (AMD)Using Rheopheresis
Brief Title: Safety and Effectiveness Investigation for Dry, Non-Exudative Age Related Macular Degeneration (AMD) Using Rheopheresis
Acronym: RHEO-AMD
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: In light of the company's current financial position we have indefinately suspended the Rheo-AMD trial.
Sponsor: OccuLogix (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RHEO-AMD 01-06
Record Dates: First submitted 2007-04-16; First posted 2007-04-17 (Estimated); Last update posted 2007-11-07 (Estimated); Status verified 2007-04

CONDITIONS: Age-Related Maculopathy
Keywords: non-Exudative (Dry) Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Rheopheresis treatment
  Interventions: Device: Rheopheresis
- 2 (Sham Comparator): Sham treatment
  Interventions: Device: Rheopheresis

INTERVENTIONS:
Device: Rheopheresis — 8 rheopheresis treatments over 10 wks.
  Arms: 1
Device: Rheopheresis — Sham treatment
  Arms: 2

SUMMARY:
SUMMARY

Age-related macular degeneration (AMD) is the leading cause of late onset visual impairment and legal blindness in people 65 years of age or older in the United States. It is a heterogeneous clinical entity in which retinal degeneration occurs predominantly in the macula in the context of aging and leads to impairment primarily of central visual acuity. The degenerative retinal eye disease occurs in two forms - a non-exudative "dry" form and an exudative "wet" form which in an individual patient may also represent stages of the disease. Non-exudative AMD accounts for 80-90% of AMD cases and it involves a constellation of clinical features that can include drusen, pigment clumping and/or retinal pigment epithelium (RPE) dropout, and geographic atrophy. Because of the overwhelming numbers of "dry" AMD subjects, the cumulative impact of this vision loss is significant.

There is no effective therapy for maintaining or improving vision associated with dry AMD. The only therapy for persons with dry AMD is an oral supplement containing high doses of antioxidants and zinc, which was tested by the National Eye Institute in a large, multi-center, double-masked, sham-controlled clinical trial1. This antioxidant therapy was shown to modestly retard the progression of dry AMD from an intermediate stage to the advanced stages and confirmed the benefit of antioxidant therapy in this disease. There is currently no FDA-approved therapy for the treatment of subjects with dry AMD.

Recently, the MIRA-1 modified per protocol population showed the effectiveness of Rheopheresis which is an application of selective therapeutic apheresis, namely double filtration plasmapheresis (DFPP) using a specifically designed filter for plasma filtration in subjects with non-exudative AMD. At one year the study reported with statistical significance (1) approximately a one line vision improvement in the Rheopheresis group versus no change in the Sham group and (2) 28% of subjects randomized to the active treatment gaining at least one line vision versus only 9% of subjects randomized to the sham treatment.

With a total of 300 subjects with dry AMD and visual acuity of 20/40-20/100 inclusive, the current investigation plans to prove the effectiveness of the Rheopheresis treatment on a larger scale. Each subject will receive a series of 8 treatments (either active treatment or sham treatment in a 2:1 ratio) for a period of approximately 2.5 months. In addition, a post-treatment ophthalmic evaluation will be performed 2 weeks after the 8th treatment (approximately 3 months after the baseline visit) and at the 6, 9 and 12 month visits. Comparing the one-year proportions of at least a 10-letter gain in ETDRS LogMar BCVA from baseline, the current investigation will show the effectiveness of Rheopheresis treatment (compared to sham treatment) for treating dry AMD subjects. Other secondary effectiveness endpoints, including mean changes and proportions of BCVA better than 20/40 at one year, will be analyzed to support the main investigation.

ELIGIBILITY:
Inclusion Criteria:

* Study eye must have a diagnosis of non-exudative, "Dry", AMD with equivalent drusen surface area of approximately 31,000 µm2 [e.g. at least 10 soft, semi-soft intermediate size ≥63µm or at least 3 drusen size ≥125 µm within 3,000 µm of the fovea documented on macular exam, retinal angiography and fundus photographs as determined by the reading center. ETDRS BCVA of 20/40 - 20/100 inclusive

Exclusion Criteria:

* Either eye with previous or active sub-retinal neovascularization (SRNV) or choroidal neovascularization (CNV)
* Pigment epithelial detachment (PED) within 500 µm of the fovea
* Either eye with a diagnosis of exudative (wet) AMD
* Subjects having undergone cataract surgery less than 3 months prior to enrollment without an open posterior capsule
* Uncontrolled hypertension and/or diabetes
* Subjects with prolonged PT/PTT (unless the subject is taking warfarin), hematocrit <35%, evidence of active bleeding, platelet count <100,000/ml

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Estimated)
Dates: Start 2007-01; Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
BCVA (Best Corrected Visual Acuity) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nozhat Choudry, PhD, Study Director — OccuLogix, Inc.
Locations (38):
- United States (32):
  - Retinal Consultants of Arizona, Phoenix, Arizona
  - Associated Retina Consultants, LTD., Phoenix, Arizona
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic, Department of Ophthalmology, Scottsdale, Arizona
  - Southwest Kidney Institute, PLC, 2149 East Warner Rd. Ste. 109 & 110, Tempe, Arizona
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Good Samaritan Hospital, Los Angeles, California
  - DSI, Brandon, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Retina Group of Washington, Chevy Chase, Maryland
  - Vitreo-Retinal Associates, Worcester, Massachusetts
  - University of Massachuesettes Medical Health Center, Worcester, Massachusetts
  - Retinovitreous Associates, Ltd., Cherry Hill, New Jersey
  - Ophthalmic Consultants of Long Island, Lynbrook, New York
  - New York Blood Center, New York, New York
  - Macula Care, New York, New York
  - Vitreous Retina Macula Consultants, New York, New York
  - Columbia University, New York, New York
  - Retina Associates of Cleveland, Beachwood, Ohio
  - Cleveland Clinic Foundation, Cole Eye Institute, Cleveland, Ohio
  - The Cleveland Clinic, Cleveland, Ohio
  - Retina Associates of Cleveland, Lakewood, Ohio
  - University of Pennsylvannia Medical Center, Philadelphia, Pennsylvania
  - Texas Retina Associates, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Memorial Hermann University of Texas Health Science Center, Houston, Texas
  - The Methodist Hospital System, Houston, Texas
  - Vitreoretinal Consultants, Houston, Texas
  - Fairfax Pathology Associates, Ltd., Annadale, Virginia
  - Retina Group of Washington, Fairfax, Virginia
- Canada (4):
  - Capital Health Systems, Ophthalmology & Visual Sciences, Halifax, Nova Scotia
  - Victoria General Hospital, Halifax, Nova Scotia
  - eyeMD Institute, Brampton, Ontario
  - Dr. Sapir, Oakville, Ontario
- Germany (2):
  - Rheopheresis Center Cologne, Cologne
  - University of Cologne, Cologne